CLINICAL TRIAL: NCT01139749
Title: Clinical, Laboratorial and Quality of Life Trial to Evaluate the Efficacy and Safety of Low-dose Oral Isotretinoin for Seborrhea.
Brief Title: Efficacy and Safety of Low-dose Oral Isotretinoin for Seborrhea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Edileia Bagatin, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: seb2010
Record Dates: First submitted 2010-06-01; First posted 2010-06-09 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Seborrhea; Seborrheic Dermatitis; Quality of Life
Keywords: oral isotretinoin; sebaceous secretion; seborrhea; seborrheic dermatitis; quality of life; Malassezia
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Isotretinoin; Salicylic Acid; Ciclopirox

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral isotretinoin (Active Comparator): Subjects from treatment arm will be treated with low-dose oral isotretinoin - 20 mg a day, every other day, for six months
  Interventions: Drug: oral isotretinoin
- salicylic acid and ciclopirox olamine (Active Comparator): Subjects from comparison arm will be treated with topical salicylic acid and ciclopirox olamine shampoo
  Interventions: Drug: salicylic acid and ciclopirox olamine

INTERVENTIONS:
Drug: oral isotretinoin — capsules of 20 mg a day, every other day, for six months
  Other Names: low-dose oral isotretinoin; off label use of oral isotretinoin
  Arms: Oral isotretinoin
Drug: salicylic acid and ciclopirox olamine — Topical salicylic acid and ciclopirox olamine shampoo for scalp and face cleansing, every other day, for six months
  Other Names: anti-seborrheic treatment; anti-dandruff treatment
  Arms: salicylic acid and ciclopirox olamine

SUMMARY:
Oral isotretinoin is the gold standard drug to treat moderate to severe acne. Other indications like seborrhea, seborrheic dermatitis have been suggested. There is risk of reversible mucocutaneous side effects, as well as alterations in lipid profile and transaminases. The major problem is teratogenicity which demands pregnancy control from treatment beginning to one month after treatment end. Seborrhea and seborrheic dermatitis are chronic conditions characterized by oily skin, hair and scalp, erythema, desquamation and negative impact on quality of life. This will be an interventional, therapeutic and quality of life randomized, comparative (parallel groups), blinded evaluation clinical trial, comprising 50 men and women, aged 18 to 40. Treatment with low-dose oral isotretinoin will be compared to topical anti-seborrheic products to evaluate the reduction of sebaceous secretion and colonization of affected areas by yeasts of Malassezia gender. Efficacy will be evaluated by clinical parameters, as well as by sebum secretion measure and application of quality of life questionnaires. Safety will be evaluated by skin hydration measure, side effects report and observation. For subjects using oral isotretinoin blood counting, transaminases, lipid profile and pregnancy test will be requested as selection criteria, on days 30 and 180. Data will be submitted to statistical analysis.

DETAILED DESCRIPTION:
Oral isotretinoin is a retinoid that controls gene expression related to cellular proliferation, differentiation, with specific action over sebocytes, reducting sebaceous gland size and secretion rate. Its binding to specific retinoid nuclear receptors is weak. It is the gold standard drug to treat moderate to severe acne. Other indications have been suggested: seborrhea, seborrheic dermatitis, rosacea and non-melanoma skin cancer prevention. There are well known reversible side effects like the mucocutaneous - cheilitis, dryness of skin, nose and eyes and risk of alterations in lipid profile and transaminases. The major problem is teratogenicity which demands pregnancy control by two different methods, from treatment beginning to one month after treatment end.

Seborrhea and seborrheic dermatitis are chronic and correlated conditions characterized by oily skin, hair and scalp, erythema, desquamation and negative impact on quality of life. Seborrhea is a very common problem, affecting 30% of population. Seborrheic dermatitis affects 3 to 5% of world population, with no differences for gender and race. The etiopathogenic factors involved in these conditions are: individual susceptibility, elevated sebaceous secretion and irritant action of products from lipophilic yeasts of Malassezia gender. The treatment usually involves topical use of corticosteroids, salicylic acid, ketoconazole, ciclopirox olamine, pimecrolimus and tacrolimus. The dermatosis impact on quality of life has been more and more evaluated by generic and specific questionnaires. The most used generic questionnaires are:"Dermatology Life Quality Index or DLQI" and "Medical Outcomes Study 36-Item Short-Form Health Survey or SF-36". Recently a specific questionnaire for oily skin named "Oily Skin Self-Image Questionnaire or OSSIQ" was published. This will be an interventional, therapeutic and quality of life randomized, comparative (parallel groups), blinded evaluation clinical trial, comprising 50 men and women, aged 18 to 40. Treatment with low-dose oral isotretinoin (20 mg a day, every other day) will be compared to topical anti-seborrheic products to evaluate the reduction of sebaceous secretion and colonization of affected areas by saprophyte yeasts of Malassezia gender. Efficacy will be evaluated by clinical parameters, as well as by sebum measure and application of two quality of life questionnaires: SF-36 and OSSIQ (after translation and validation for Brazilian Portuguese). Safety will be evaluated by skin hydration measure, side effects report and observation. The devices Sebumeter and Corneometer, from Courage & Khazaka, Köln, Germain, will be used. For subjects using oral isotretinoin blood counting, transaminases, lipid profile and pregnancy test will be requested as selection criteria, on days 30 and 180. Results will be submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* consent form signature
* presence of seborrhea and / or seborrheic dermatitis on face and scalp
* good health
* no previous treatment with oral isotretinoin in the last 6 months
* normal laboratorial tests: pregnancy test, blood counting, transaminases and lipide profile
* concordance on use of two anticonceptional methods, during and until one month after the end of the study

Exclusion Criteria:

* difficulty to follow study conditions
* pregnancy risk
* diabetes
* collagen diseases
* bone or muscles diseases
* alcohol abuse
* hypervitaminosis A

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Sebum secretion rate | day 0
  Sebum secretion measure on forhead, along scalp line, using Sebumeter,Courage & Khazaka, Köln, Germany.
sebum secretion rate | day 180
  Sebum secretion measure on forhead, along scalp line, using Sebumeter, Courage & Khazaka, Köln, Germany

SECONDARY OUTCOMES:
Oral isotretinoin side effects | day 0
  Laboratorial tests for oral isotretinoin side effects evaluation: pregnancy test, blood counting, transaminases and lipide profile
oral isotretinoin side effects | day 30
  Laboratorial tests for oral isotretinoin side effects evaluation: pregnancy test, blood counting, transaminases and lipide profile
oral isotretinoin side effects | day 180
  Laboratorial tests for oral isotretinoin side effects evaluation: pregnancy test, blood counting, transaminases and lipide profile

CONTACTS AND LOCATIONS:
Overall Officials: Edileia Bagatin, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo - Dermatology Department - Cosmetic Dermatology Unit, São Paulo, São Paulo, Brazil